CLINICAL TRIAL: NCT03314337
Title: A Prospective Randomized Controlled Study Comparing Outcomes of Distal Pancreatectomy With or Without Pancreatic Stent
Brief Title: Pancreatic Stent for Distal Pancreatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Weishen WANG, doctor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HBP-RCT-002
Record Dates: First submitted 2017-10-06; First posted 2017-10-19 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Distal Pancreatectomy
Keywords: Distal Pancreatectomy; Pancreatic stent; Post-operative pancreatic fistula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distal Pancreatectomy without pancreatic stent (No Intervention)
- Distal Pancreatectomy with pancreatic stent (Experimental): pancreatic stent will be placed in the main pancreatic duct during the operation
  Interventions: Device: Pancreatic stent: PSOF COOK®

INTERVENTIONS:
Device: Pancreatic stent: PSOF COOK® — After removing the distal pancreas, PSOF COOK will be place in the main pancreatic duct
  Arms: Distal Pancreatectomy with pancreatic stent

SUMMARY:
The purpose of this study is to compare outcomes of patients undergoing distal pancreatectomy with or without pancreatic stent

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing distal pancreatectomy
2. Signed the informed consents

Exclusion Criteria:

1. Recurrence patients
2. pre-operative anti-cancer treatment
3. patients with contraindication(hepatic/ respiratory/ renal dysfunction, etc )
4. AJCC stage IV
5. pre operative oddi'ssphincter incision
6. operation non radical
7. pancreatic stent not at place

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
all-cause mortality / complications | Hospitalization 30days（duration of hospital stay)
  mortality, pancreatic fistula, Biliary fistula，bleeding， etc

SECONDARY OUTCOMES:
all-cause mortality / complications | 30 days after operation
  mortality, pancreatic fistula, Biliary fistula，bleeding， etc

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided